CLINICAL TRIAL: NCT05011097
Title: A Phase I Study to Evaluate the Safety, Tolerability, PK/PD and Immunogenicity Characteristics of Recombinant Anti-CD38 and Anti-CD3 Bispecific Antibodies (Y150) for Injection in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Phase I Clinical Trial of Y150 in the Treatment of Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wuhan YZY Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y15001
Record Dates: First submitted 2021-07-15; First posted 2021-08-18 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Y150 (Experimental): Subjects who meet the enrollment criteria will enter the core treatment period and receive a cycle of treatment with Y150 (once weekly for 4 weeks) via intravenous infusion. And eligible subjects who complete the core treatment period will receive a cycle of extended treatment (once weekly for 4 weeks) until disease progression or toxicity intolerance.
  Interventions: Drug: Y150

INTERVENTIONS:
Drug: Y150 — Subjects will receive an intravenous infusion of Y150 in a dose escalation once a week for a 28-day treatment cycle until confirmed progression, unaccepted toxicity, or any criterion for withdrawal from the study.

SUMMARY:
The main purpose of this Phase I study is to access the safety and tolerability of Y150 at different dose levels. It is hoped to find out the recommended dose for Phase II/III.

DETAILED DESCRIPTION:
This is a Phase I, open-label，dose-escalation trial in patients with relapsed or refractory multiple myeloma. There are two parts of the study: a dose-escalation part and a dose-expansion part. Dose escalation follows an accelerated design initially with 2 single subject cohorts (Cohorts 1-2) and switches to a classical 3+3 design (Cohorts 3-7). Dose-expansion means that at least 9 subjects (included subjects of the dose-escalation part) will be selected in 1 - 3 dose levels to focus on the pharmacokinetics (PK) / pharmacodynamic (PD) features and recommended dose for Phase II (RP2D). Additional purpose of the study is to find out whether the study drug has anti-tumor effects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years.
2. Subject has a history of multiple myeloma with relapsed and refractory disease, and must have received at least 2 prior multiple myeloma treatment regimens (including a proteasome inhibitor and an immunomodulatory agent), or can not tolerate the toxicity of PIs and IMIDS; or have drug resistance to one and toxic intolerance to the other.

   1. Relapsed multiple myeloma is defined as IMWG criteria in 2016, including clinical relapse or relapse after CR.
   2. Refractory multiple myeloma is defined as failure of initial or salvage therapy to achieve at least a minimal response (only achieve SD after treatment ≥ 2 cycles ), or disease progression during treatment or within 60 days after the last treatment.
3. Subjects must have measurable disease, including at least one of the criteria below:

   1. M-protein ≥ 10 g/L by SPEP/immunofixation for subjects with immunoglobulin class G (IgG) myeloma , M-protein ≥ 5g/L for subjects with IgA, IgD, IgE, IgM myeloma or
   2. ≥ 200 mg/24 hours urine collection by UPEP or
   3. Serum free light chain (FLC) levels ≥ 100 mg/L and an abnormal kappa/lambda (κ/λ) ratio in patients without detectable serum or urine M-protein
4. The interval between the last anti-tumor treatment and the first administration of Y150 (including PIS and IMADs) ≥4 weeks, the interval between CD38 mAb administration and the first administration of Y150 ≥12 weeks;
5. ECOG performance status 0 - 2;
6. Life expectancy ≥ 3 months
7. Adequate hematological function as evidenced by meeting all the following requirements:

   1. Absolute neutrophil count ≥1.0×109/L (growth factor support not allowed within 48h)
   2. Hemoglobin > 70 g/L( without blood transfusion within 7 days)
   3. Platelet count ≥50×109/L(without transfusion within 7 days)
8. Adequate hepatic function as evidenced by meeting all the following requirements:

   1. Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
   2. Aspartate aminotransferase (AST), and alanine aminotransferase (ALT)≤ 2.5 × ULN;
9. Calculated creatinine clearance (CrCL) ≥ 30 mL/min
10. Understand and voluntarily sign written informed consent.

Exclusion Criteria:

1. Subject has central nervous system involvement of multiple myeloma.
2. Subject has received ≥ 10 mg/day prednisone equivalent within one week before starting Y150.
3. Subject with primary or secondary plasma cell leukemia.
4. Subject had a prior autologous stem cell transplant ≤ 12 weeks months prior to starting Y150, or had a prior autologous stem cell transplant history.
5. Subject received a chimeric antigen receptor T (CAR T) cell product ≤ 6 months prior to starting Y150.
6. Concurrent malignancy within 5 years prior to entry other than adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin, basal cell carcinoma, prostate cancer under active surveillance, prostate cancer that has undergone definitive treatment, ductal carcinoma in situ of the breast, or ≤ T1 urothelial carcinoma.
7. Allergy to Abs drugs or human protein.
8. Active infection(CTCAE Grade ≥2).
9. Subjects with severe respiratory disease, and to be unsuitable to participate in study by investigators judgment.
10. Severe cardiovascular disease, including a history of CABG or PCI, myocardial infarction within 6 months of study entry, unstable angina ,NYHA class III or IV heart failure, uncontrolled hypertension or left ventricular ejection fraction <50%
11. QTc interval > 480 ms; Family or personal with a history of long or short QT syndrome; significant clinical history of ventricular arrhythmias, or currently receiving antiarrhythmic drugs or implanted defibrillator to treat ventricular arrhythmias.
12. Patients with a history of active autoimmune diseases (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis etc.), except when the disease is in a stable state (without systemic immunosuppressant treatment, the symptoms are stable for more than 6 months).
13. Patients with severe hyperthyroidism or hypothyroidism.
14. Patients with metabolic diseases such as uncontrolled diabetes, severe gastrointestinal bleeding, severe diarrhea (Grade ≥ 2 according to CTCAE), or severe gastrointestinal obstruction requiring intervention.
15. Patients with a history of immunodeficiency, including HIV positive.
16. HIV antibody, TP antibody and HCV antibody were positive, HBsAg positive and hepatitis B virus DNA test showed that patients with active hepatitis B (HBV-DNA ≥ 1000cps/ml).
17. Patients who have received inoculation of (attenuated) live virus vaccine within 4 weeks before the first administration.
18. Pregnant, lactating women, or females or males who have fertility plan within 6 months during the study and after the end of the medication.
19. Patients with a previous history of definite neurological or psychiatric disorders, and investigator believe that it affects patients' cognitive function or compliance, including unstable epilepsy, dementia, schizophrenia, etc.
20. Any condition that the investigator believes may not be appropriate for participating the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events according to CTCAE V5.0 | up to approximately 2 years
  An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Number of Participants With Dose Limiting Toxicities (DLTs) | From the time of first dosing (Day 1) until the forth dosing (Day 28)
  DLTs were assessed using the national cancer institute common terminology criteria for adverse events (NCI-CTCAE) version 5.0.

SECONDARY OUTCOMES:
Area under the curve (AUC) of Y150 | Up to 1 weeks after the fourth dosing.
Peak Plasma Concentration (Cmax) of Y150 | Up to 1 weeks after the fourth dosing.
Half-time (t1/2) of Y150 | Up to 1 weeks after the fourth dosing.
lymphocyte subsets in peripheral blood | 12 months (anticipated)
  including CD3/CD4/CD8/CD14/CD19/CD38/CD45/CD56/CD69 lymphocyte subsets in peripheral blood
Cytokines levels in serum | 12 months (anticipated)
  including IL-2, IL-6, IL-8, IL-10, TNF-α, IFN-α, IFN-γ levels in serum
Anti-drug antibodies(ADAs) titer | 12 months (anticipated)
neutralizing antibody titer | 12 months (anticipated)
Objective Response Rate (ORR) | 12 months (anticipated)
  ORR is defined as percentage of participants who achieved stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR), based on International Myeloma Working Group (IMWG) criteria.
Time to Progression (TTP) | 12 months (anticipated)
  TTP was defined as the number of days from the date of first infusion (Day 1) to the date of first record of disease progression.
Duration of Response | 12 months (anticipated)
  Duration of response was calculated from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the International Myeloma Working Group (IMWG) criteria.
Progression-Free Survival (PFS) | 12 months (anticipated)
  PFS was defined as the time between the date of first dose of Y150 and either disease progression or death, whichever occurs first.
Overall Survival (OS) | 12 months (anticipated)
  OS was defined as the number of days from administration of the first infusion (Day 1) to date of death.
Time to first Response | 12 months (anticipated)
  Time to first response was defined as the time from the date of first dose of Y150 to the date of initial documentation of a response (PR or better).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No